CLINICAL TRIAL: NCT01901601
Title: Randomized Clinical Trial of OCT-Guided Laser-Assisted Lamellar Anterior Keratoplasty in Adults for Stromal Opacities
Brief Title: LALAK for Opacities
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Modifying procedure.
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Winston Chamberlain, MD, PhD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB#00009282; R01EY018184 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: STROMAL OPACITIES
Keywords: KERATOPLASTY; STROMAL OPACITIES
MeSH Terms: interventions — Anesthesia, General; Tomography, Optical Coherence; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LALAK (Experimental): laser-assisted lamellar anterior keratoplasty. Optical Coherence Tomography, femtosecond laser, topical anesthesia, and Retrobulbar Block or General Anesthesia will be used.
  Interventions: Procedure: LALAK; Drug: Retrobulbar Block or General Anesthesia; Device: optical coherence tomography (OCT); Drug: Topical Anesthesia; Device: femtosecond laser
- IEK (Active Comparator): Intralase-enabled keratoplasty. Femtosecond laser and Retrobulbar Block or General Anesthesia will be used.
  Interventions: Procedure: IEK; Drug: Retrobulbar Block or General Anesthesia; Device: femtosecond laser

INTERVENTIONS:
Procedure: LALAK — 1. A "dovetail" shaped cut will be made on the graft using a femtosecond laser at the eye bank. The cut depth will be proportional to the central stromal thickness of the graft. This graft will be separated from stromal bed by eye bank personnel for examination of the cut surface. High-quality graft will be replaced in preservation medium and shipped to the surgeon prior to surgery.
  2. The host cornea will receive femtosecond laser cut consisting of a shallow lamellar cut with angled side cut to match the dovetail graft in a tongue-in-groove fashion. The femtosecond laser treatments will be performed under topical anesthesia in the laser suite. The femtosecond laser is an FDA-approved device for use in this indication (corneal transplantation including lamellar keratoplasty). A protective eye shield is placed over the eye. The graft will be sutured into the host bed.
  Arms: LALAK
Procedure: IEK — 1. A full thickness graft will be prepared at the eye bank with zigzag side cuts prepared with a femtosecond laser. The graft is separated from the rim, replaced in the preservation medium, and shipped to the surgeon prior to the surgery.
  2. In the laser suite, the host cornea will be cut with the femtosecond laser with zigzag side cuts leaving a 70-100 micron bridge. A protective eye shield is placed over the eye. The graft will be sutured into the host bed.
  Arms: IEK
Drug: Retrobulbar Block or General Anesthesia
Device: optical coherence tomography (OCT) — OCT will be used to guide the depth of the graft and donor dissections. The OCT systems to be used in this study will be the RTVue (Optovue, Inc., Fremont, CA) or the Visante (Carl Zeiss Meditec, Inc., Dublin, CA). Both are FDA-approved for the mapping of corneal thickness.
  Arms: LALAK
Drug: Topical Anesthesia
  Arms: LALAK
Device: femtosecond laser — The femtosecond laser system to be used in this study for host cornea preparation will be the Intralase FS system (iFS, AMO, Inc., Santa Ana, CA). The iFS is FDA-approved for corneal surgery including full thickness and lamellar keratoplasty. Eye banks use earlier versions of the Intralase system which are also FDA approved for this indication.

SUMMARY:
The purpose of this protocol is to compare and develop new surgical technique of partial-thickness corneal transplantation for treating corneal opacity. A newly developed technique, "dovetail" laser-assisted lamellar anterior keratoplasty (LALAK), will be tested and compared with standard full-thickness corneal transplantation, Intralase-enabled keratoplasty (IEK). The new LALAK technique replaces only the front portion of the cornea and does not have the risks associated with conventional IEK. Additionally, optical coherence tomography (OCT) will be used to guide the depth of the graft and donor dissections.

The data will be analyzed to understand whether the new technique (LALAK) can repeatedly achieve good visual outcomes with lower risk from the operation compared to the visual outcomes and risk associated with the current standard of care, IEK.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with corneal opacities that cannot be adequately or safely corrected with spectacles, contact lens or excimer laser surface ablation. The cornea must have healthy endothelium (endothelial cell density > 1,500/mm2).

Exclusion Criteria:

1. Preoperative corneal thickness less than 400 microns.
2. Inability to give informed consent.
3. Corneal edema
4. Central guttata
5. Inability to maintain stable fixation for OCT imaging.
6. Inability to commit to required visits to complete the study.
7. Eyes with concurrent cataract, retinal diseases, glaucoma, or other eye conditions that may limit the visual outcome after surgery.
8. Patients with severe collagen vascular diseases or ocular surface disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
BSCVA (Snellen chart) | 24 months
  A primary outcome measures will be BSCVA (Snellen chart)
intraoperative perforation rate | 24 months
  A primary outcome measure will be intraoperative perforation rate.

SECONDARY OUTCOMES:
postoperative refractive error | 24 months
  A secondary outcome measures will be postoperative refractive error
topographic astigmatism | 24 months
  A secondary outcome measures will be topographic astigmatism
interface clarity | 24 months
  A secondary outcome measures will be interface clarity (masked OCT and confocal microscopy grading)
endothelial cell count | 24 months
  A secondary outcome measures will be endothelial cell count (specular microscopy)
complications | 24 months
  A secondary outcome measures will be complications (rejection, interface opacification, others).

CONTACTS AND LOCATIONS:
Overall Officials: Winston Chamberlain, MD, PhD, Principal Investigator — Casey Eye Institute, Oregon Health & Science University

REFERENCES:
- See also: Related Info — http://www.coollab.net